CLINICAL TRIAL: NCT01453647
Title: Self-Efficacy, Stress, Immunity and Symptoms of Fibromyalgia
Brief Title: Study to Explore the Relationships Among Immunity and Stress and the Symptoms of Fatigue, Pain, and Mood Following Guided Imagery in Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12211
Record Dates: First submitted 2011-08-12; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; self-efficacy; fatigue; stress; cytokine
MeSH Terms: conditions — Fibromyalgia; Fatigue | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guided Imagery (Experimental): The intervention consists of three audio-recorded guided imagery scripts formatted as three separate tracks on one CD. Each track is 30 minutes in length and is to be used in a recommended order for the first 6 weeks of the intervention and then used in any order for the follow-up weeks, 7 through 10. Project participants will be instructed to use each CD track, as prescribed, a minimum of once daily. CD Track 1 is a basic relaxation entrainment script; CD track 2 is a pleasant scene imagery script; CD track 3 is a well body imagery script.
  Interventions: Other: Guided Imagery
- control (No Intervention): Participants in the control group will be instructed to maintain their FM treatment regimens as reported at baseline.

INTERVENTIONS:
Other: Guided Imagery — The intervention consists of three audio-recorded guided imagery scripts formatted as three separate tracks on one CD. Each track is 30 minutes in length and is to be used in a recommended order for the first 6 weeks of the intervention and then used in any order for the follow-up weeks, 7 through 10. Project participants will be instructed to use each CD track, as prescribed, a minimum of once daily. CD Track 1 is a basic relaxation entrainment script; CD track 2 is a pleasant scene imagery script; CD track 3 is a well body imagery script.
  Arms: Guided Imagery

SUMMARY:
This project will be the first known to explore the relationships among immunity and stress and the symptoms of fatigue, pain, and mood following guided imagery in women with fibromyalgia. Finding ways to reduce these unpleasant symptoms may lead to improved function and well-being in this chronic disorder.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic widespread pain and fatigue syndrome that affects 3 to 6 million adults in the United States. Consequences of FM include physical and psychological distress, loss of work productivity, reduced quality of life, and increased use of health resources. Although the mechanisms underlying the symptomatology of FM are not clear; one theory suggests potential alterations in cytokine balance. Because the symptoms of FM may be worsened by stress and negative psychological processes, mind-body modalities may positively influence the neuroendocrine and immunological mediators of symptoms in FM. Given that immune modulation by both psychosocial stressors and interventions has been linked to health changes, self-efficacy (i.e., the belief that one can cope), may be one mechanism affecting FM outcomes. The specific aims of this project are: (1) to test the effects of a 10-week guided imagery intervention in comparison to an attention control group among women diagnosed with fibromyalgia on (a) the primary outcomes of self-efficacy for managing symptoms and perceived stress and (b) the secondary outcomes of symptoms of fatigue, pain, distressed mood, and depressive symptoms and markers of immune function; and (2) to examine the relationships among self-efficacy for managing symptoms, perceived stress, symptoms of fatigue, pain, distressed mood, and depressive symptoms and markers of immune function. The biobehavioral framework to guide this project is adapted from psychoneuroimmunology. Using a randomized controlled two-group design with repeated measures, 72 individuals will be recruited and randomized into one of two groups: Usual Care plus guided imagery (GI) intervention (Group 1) or Usual Care alone (i.e., attention control group) (Group 2). The intervention consists of three 30-minute guided imagery audio recordings to be used in a proscribed manner over a 10-week period. An ANCOVA model will be used to test for group differences between the intervention and standard care groups at week 10. This project will be the first known to explore the relationships among cytokines and perceived stress and the symptoms of fatigue, pain and mood following the administration of a biobehavioral intervention in women with FM.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and older
* female
* diagnosis of FM based on the American College of Rheumatology criteria and documented by the patient's primary physician
* no known major psychiatric or neurological conditions that would interfere with project participation
* able to speak and read standard English
* a minimum of a 6th grade education level
* an ability to understand and sign the consent form and understand and complete the pencil and paper assignments

Exclusion Criteria:

* presence of other systemic rheumatologic conditions such as rheumatoid arthritis, systemic lupus erythematosus, and/or Sjogren's Disease
* history of epilepsy
* any present psychiatric disorder involving a history of psychosis (e.g., schizophrenia, schizoaffective disorder; schizophreniform disorder, delusional disorder, etc.)
* being immunocompromised
* receiving corticosteroid treatments
* being pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Fatigue | baseline
  Measured by Multidimensional Fatigue Symptom Inventory-Short Form(MFSI-SF), PROMIS Fatigue Short-Form, and Brief Fatigue Invebtory (BFI) and 17 cytokines
Fatigue | 6th weeks
  Measured by Multidimensional Fatigue Symptom Inventory-Short Form(MFSI-SF), PROMIS Fatigue Short-Form, and Brief Fatigue Invebtory (BFI) and 17 cytokines
Fatigue | 10th week
  Measured by Multidimensional Fatigue Symptom Inventory-Short Form(MFSI-SF), PROMIS Fatigue Short-Form, and Brief Fatigue Invebtory (BFI) and 17 cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Menzies, PhD, APRN-BC, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Common Wealth University Health System, Richmond, Virginia, United States